CLINICAL TRIAL: NCT06305286
Title: A Pilot Study Assessing the Safety of Using a Monoclonal Antibody Against Cluster of Differentiation 40 (CD40) Ligand to Achieve a Calcineurin Inhibitor-free Immunosuppression Regimen in Patients With Type 1 Diabetes Mellitus (T1D) and Problematic Hypoglycemia Undergoing Islet Cell Transplantation
Brief Title: Safety, Tolerability, and Efficacy of Immunomodulation With A Monoclonal Antibody Against CD40L in Combination With Transplanted Islet Cells in Adults With Brittle Type 1 Diabetes Mellitus (T1D)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Cure Alliance (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB23-1367
Record Dates: First submitted 2024-02-16; First posted 2024-03-12 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: AT-1501 — AT-1501 is a monoclonal antibody for Injection is a humanized immunoglobulin G1 (IgG1) kappa monoclonal anti-CD40L antibody that blocks CD40L binding to its receptor, CD40.

SUMMARY:
AT-1501 is a monoclonal antibody. Antibodies are Y-shaped proteins that are produced naturally by the subject's immune system to attack and fight foreign substances that cause illness. Monoclonal antibodies are man-made proteins manufactured to serve as substitute antibodies to fight diseases. Monoclonal antibodies can restore, enhance, or mimic (copy) the immune system's attack process; they can also tone down the immune system. AT-1501 is thought to work by dampening down the immune system so that it will be less likely to attack the transplanted cells. For other types of transplants, like kidney, a drug called a calcineurin inhibitor is usually used to prevent rejection. That class of drugs can be toxic to islet cells. AT-1501 is an experimental agent that is anticipated to prevent rejection without harming the islet cells.

DETAILED DESCRIPTION:
By doing this study, the study team is studying an investigational regimen containing 2 experimental components:

* An investigational drug called AT-1501 and
* Human pancreatic islet cells

Both AT-1501 and human pancreatic islet cells are considered investigational because they are not currently approved for use in the United States.

Islet cells are the specialized cells in the pancreas that produce insulin. In this study, islet cells will be collected from the pancreas of a deceased organ donor and transplanted into the body. The goal of this study is to see whether these transplanted islet cells can take over insulin production. The study team will evaluate how well the subject makes insulin and how well-controlled blood sugar is after the transplant.

The islet transplant procedure involves inserting a thin, flexible tube called a catheter through a small cut in the upper abdomen. A radiologist uses X-rays and ultrasound to guide the catheter into the portal vein of the liver where the islet cells are delivered. This study of islet transplantation will test to see if islet transplantation is safe and effective.

Because these islet cells come from another person, the subject's immune system may recognize them as foreign and attack them. Standard immunosuppressive medicines (Anti-thymocyte globulin [ATG] or Basiliximab, mycophenolate mofetil/mycophenolate sodium (MMF/MPS) (CellCept®), and Etanercept) will be used to help prevent the body from attacking the transplanted islet cells. AT-1501 will be given in combination with these standard immunosuppressive medicines to test whether the investigational drug is safe, tolerable, and efficacious. The effect of the combination of AT-1501 with other immunosuppressant medications has not been previously tested.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 18-65 years of age.
2. A diagnosis of T1D ≥5 years with onset of disease at <40 years of age.
3. Ability to provide informed consent.
4. Able to comply with study procedures, including the requirement to utilize continuous glucose monitoring (CGM).
5. Involvement in appropriate diabetes management in accordance with the standard of care, as directed by an endocrinologist or diabetologist with at least 4 (quarterly) clinical evaluations within the 12 months prior to Screening; using CGM*: using an insulin pump or multiple daily injection (MDI) of insulin therapy; and, unable to achieve acceptable metabolic control because of the occurrence of unexplained SHEs- at least 3 unexplained SHEs not secondary to a missed meal or dosing error, in the 12 months prior to Screening.

   *CGM will be provide to subjects who otherwise qualify for study participation but have not used CGM previously.
6. At least 3 unexplained SHEs not secondary to a missed meal or dosing error, in the 12 months prior to Screening.
7. HbA1c level 7.0% (48 mmol/mol) to 9.5% (80 mmol/mol), inclusive.
8. Absence of stimulated C-peptide (<0.3 ng/mL) in response to a 240-minute mixed- meal tolerance test (MMTT).
9. Impaired awareness of hypoglycemia (IAH) as defined by a Clarke Score [Clarke 1995] of 4 or more at the time of Screening, during the Screening period, and within the last 6 months prior to the transplant.
10. If female, must be surgically sterile or 2 years postmenopausal. Women of childbearing potential may be enrolled if a serum pregnancy test is negative at screening/baseline. Women of childbearing potential and men with partners that are of childbearing potential must agree to use 2 forms of highly effective methods of contraception from Screening, throughout the study, and while receiving immunosuppressive therapy for the functioning graft after the conclusion of the study. Contraception use must continue for 90 days after the last administration of the study drug (see Appendix 5). Male participants must refrain from donating sperm for the duration of the study and agree to not donate sperm for 90 days after last administration of the study drug.
11. Patients with Coronavirus Disease 2019 (COVID-19) Polymerase chain reaction (PCR) negative test result.

Exclusion Criteria:

1. Any previous solid organ or islet allotransplant.
2. Body mass index (BMI) >30 kg/m2.
3. Weight ≤50 kg.
4. Insulin requirement >1.0 unit/kg/day or <15 units/day.
5. Treatment with any anti-diabetic medication other than insulin within 4 weeks of Screening.
6. Uncontrolled proliferative diabetic retinopathy.
7. Blood pressure: systolic blood pressure (SBP) >140 mmHg or diastolic blood pressure (DBP) >90 mmHg.
8. Estimated glomerular filtration rate (eGFR) calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation <60 mL/min/1.73 m2.
9. Diagnosis of macroalbuminuria (>300 mg/g creatinine).
10. For female participants: Positive pregnancy test, presently breast-feeding, or unwillingness to use effective contraceptive measures for the duration of the study and 90 days after discontinuation. For male participants: intent to procreate during the duration of the study or within 90 days after discontinuation or unwillingness to use effective measures of contraception.
11. History of malignancy except for completely resected squamous or basal cell carcinoma of the skin.
12. History of a thromboembolic event (TE), known hypercoagulable state, or condition requiring long-term anticoagulation.

    a. Participants with a history of clotted venous access not requiring long- term anticoagulation may be included at the Principal Investigator's discretion if they have no other history of TEs or known hypercoagulable state.
13. Known heparin allergy.
14. Receiving treatment for a medical condition requiring chronic use of systemic steroids, except for physiologic replacement for example in Addison disease.
15. Presence of ongoing active infection including tuberculosis (TB), human immunodeficiency virus (HIV), hepatitis B, hepatitis C. Laboratory evidence of active infection even in the absence of clinical symptoms of infection is exclusionary.
16. Invasive aspergillus, histoplasmosis or coccidioidomycosis infection within one year prior to Screening.
17. Negative screen for Epstein-Barr Virus (EBV) by immunoglobulin G (IgG) determination.
18. Current treatment with any immunosuppressive regimen, and treatment with biologic immune modulating agents, Janus kinase (JAK) inhibitors, sphingosine-1-phosphate (S1P) receptor agonists, azathioprine, Mercaptopurine (6- MP), or systemic corticosteroids in the previous 5 years.
19. Persistent elevation of serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) value greater than 3 times the upper limit of normal (ULN); elevation of total bilirubin >1.5 ULN.
20. Any history of receiving experimental cell or gene therapy. Exposure to any other experimental or investigational agent within 30 days or 5 half-lives; whichever is longer.
21. History of substance abuse within the past 2 years.
22. Allergy to the Boost drink necessary for MMTT
23. Severe cardiovascular disease characterized by any one of these conditions: a) stroke;

    b) recent myocardial infarction (within past 6 months); c) evidence of ischemia on functional cardiac exam within the last year; d) left ventricular ejection fraction <30%.
24. History of significant gastrointestinal disease such as symptomatic cholecystolithiasis; acute or chronic pancreatitis; symptomatic peptic ulcer disease; severe unremitting diarrhea, vomiting or other disorders potentially interfering with the ability to absorb oral medications.
25. Significant hyperlipidemia despite medical therapy defined as fasting low-density lipoprotein (LDL) cholesterol >130 mg/dL and/ or triglycerides >200 mg/dL.
26. History of any conditions that can interfere in the assessment of HbA1c due to increased red blood cell turnover or requirement for regular blood transfusions such as sickle cell disease (HbSS, hematopoietic blood stem cell (HbSC), HbS/beta thalassemia); Beta thalassemia major; Alpha Thalassemia (HbH) disease, Hemoglobin H-Constant Spring.
27. History of any other acute or chronic medical condition or pre-planned medical/surgical procedure that, in the opinion of the Principal Investigator, would compromise the safety of participants or the integrity of study results; non- compliance with recommended diabetes care in the preceding 12 months.
28. Baseline Hb below the lower limits of normal at the local laboratory; lymphopenia (<1,000/µL), neutropenia (<1,500/µL), or thrombocytopenia (platelets <100,000/µL). Participants with lymphopenia are allowed if the Principal Investigator determines there is no additional risk and obtains clearance from a hematologist.
29. Any coagulopathy or medical condition requiring long-term anticoagulant therapy (e.g., warfarin) after islet cell transplantation (low-dose aspirin treatment is allowed) or participants with an international normalized ratio (INR) >1.5. The use of Plavix is allowed only when portal vein access is obtained using a mini-laparotomy procedure at the time of islet cell transplant.
30. History of factor V deficiency.
31. Administration of live attenuated vaccine(s) within 2 months of Screening.
32. Any previous treatment with AT-1501 or any other anti-CD40L therapy
33. Baseline Panel-reactive Antibody (PRA) over 20%
34. Patients with COVID-19 positive PCR tests.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who are insulin-independent post- first and final transplant | Day 75 and Day 365

SECONDARY OUTCOMES:
Number of Participants with glycosylated hemoglobin (HbA1c) <7.0% | at Day 365

OTHER OUTCOMES:
Number of Participants with free of serious hypoglycemic events (SHEs) post-first and final transplant | Day 28 to Day 365
Number of Participants with HbA1c ≤6.5% AND free from SHEs post-first and final transplant. | at Day 365 and from Day 28 through to Day 365
Number of Participants with graft failure post final transplant. | Day 365
Number of participants with impaired awareness of hypoglycemia after final islet cell transplant and after discontinuation of AT-1501. | Day 75 and 365, 1-3 years
Change in glycemic lability after final islet cell transplant and years after discontinuation of AT-1501 | Day 75 and 365, 1-3 years
Change in albumin excretion ratio (AER) post-first and final transplant. | Day 365
Change in estimated glomerular filtration rate (eGFR) post-first and final transplant. | Day 365
Change in percent new macroalbuminuria post-first and final transplant. | Day 365
Change in variability after final islet cell transplant and years after discontinuation of AT-1501 | Day 75 and 365, 1-3 years

CONTACTS AND LOCATIONS:
Overall Officials: John Fung, MD PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No